CLINICAL TRIAL: NCT00558155
Title: Title: The Impact of Immunostimulating Nutrition on Infectious Complications After Upper Gastrointestinal Surgery - A Prospective, Randomized, Clinical Trial.
Brief Title: The Impact of Immunostimulating Nutrition on the Outcome of Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1st Dept Surg
Record Dates: First submitted 2007-11-09; First posted 2007-11-14 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Gastric Cancer; Pancreatic Cancer
Keywords: immunonutrition; enteral nutrition; parenteral nutrition; surgery
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Hyperphagia | interventions — Parenteral Nutrition; fish oil triglycerides; alanylglutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SEN (Experimental): standard enteral nutrition
  Interventions: Drug: peptisorb
- IMEN (Experimental): immunostimulating enteral nutrition
  Interventions: Drug: Stresson
- SPN (Experimental): standard parenteral nutrition
  Interventions: Drug: Parenteral nutrition
- IMPN (Experimental): immunostimulating parenteral nutrition
  Interventions: Drug: Omegaven, Dipeptiven

INTERVENTIONS:
Drug: peptisorb — standard isocaloric eteral diet (1 ml = 1 kcal)
  Arms: SEN
Drug: Stresson — Oligopeptic, enteral diet (1 ml=1.25 kcal)
  Arms: IMEN
Drug: Parenteral nutrition — Protein requirements were covered by 10 and 15% amino acid solutions (Aminoplasmal, B Braun, Poland). Energy requirements were covered by glucose (10, 20 and 40% solutions, B Braun, Poland) and lipid emulsions (10 and 20% Lipofundin MCT/ LCT, B Braun, Poland). Addtional: Tracutil, Addamel
  Arms: SPN
Drug: Omegaven, Dipeptiven — Immunostimulating components: Omegaven (omega-3-fatty acids) and Dipeptiven (Glutamine Arginine) Protein requirements were covered by 10 and 15% amino acid solutions (Aminoplasmal, B Braun, Poland). Energy requirements were covered by glucose (10, 20 and 40% solutions, B Braun, Poland) and lipid emulsions (10 and 20% Lipofundin MCT/ LCT, B Braun, Poland). Addtional: Tracutil, Addamel
  Arms: IMPN

SUMMARY:
The aim of the study was to assess the clinical effect of immunostimulatory enteral and parenteral nutrition in patients undergoing resection for gastrointestinal cancer. 205 subjects were randomly assigned into four study groups, standard and immunostimulating, enteral and parenteral. The study was designed to test the hypothesis that immunonutrition and enteral nutrition would reduce the incidence of infectious complications following upper gastrointestinal surgery.

DETAILED DESCRIPTION:
All patients qualified between June 2001 and December 2005 to total and distal subtotal gastrectomy or pancreaticoduodenectomy were screened for eligibility to participate in the study. Additional eligibility criteria included: age between 18 and 80 years, Karnofsky performance status score of 80 or more, and adequate organ function measured by routine blood tests. Patients requiring preoperative nutritional support, as well as those with disseminated tumors, serious comorbidities (American Society of Anesthesiologists risk class of 4 or 5), and renal or liver failure were excluded. The study was designed to test the hypothesis that immunonutrition and enteral nutrition would reduce the incidence of infectious complications following upper gastrointestinal surgery. Therefore, patients were randomly assigned in a 2×2 factorial design to four groups receiving immunostimulating versus normal diets, and enteral versus intravenous nutritional support. The secondary objective of the study was to evaluate the effect of nutritional intervention on overall morbidity and mortality rates, and the length of hospital stay.

After completing tumor resection, patients who met the eligibility criteria were intraoperatively assigned to either of the treatment groups using sealed envelopes containing computer-generated allocation numbers. The following groups were generated: standard enteral nutrition (SEN), immunostimulating enteral nutrition (IMEN), standard parenteral nutrition (SPN), and immunostimulating parenteral nutrition (IMPN). The study was carried out following the international ethical recommendations stated in the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* resectable gastric or pancreatic cancer
* age between 18 and 80 years,
* Karnofsky performance status score of 80 or more,
* adequate organ function

Exclusion Criteria:

* unresectable gastric or pancreatic cancer
* patients requiring preoperative nutritional support,
* disseminated tumors,
* serious comorbidities (American Society of Anesthesiologists risk class of 4 or 5),
* renal or liver failure were excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2001-06; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
During the postoperative period, all patients were observed for both surgical and non-surgical complications | 52 months

SECONDARY OUTCOMES:
The secondary objective of the study was to evaluate the effect of nutritional intervention on overall morbidity and mortality rates, and hospital stay. | 52 months

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, PhD, MD, Principal Investigator — Jagiellonian University 1 Dept Surgery
Locations (1):
- 1st Department of General Surgery, Krakow, Poland

REFERENCES:
- [Derived] Klek S, Sierzega M, Szybinski P, Szczepanek K, Scislo L, Walewska E, Kulig J. Perioperative nutrition in malnourished surgical cancer patients - a prospective, randomized, controlled clinical trial. Clin Nutr. 2011 Dec;30(6):708-13. doi: 10.1016/j.clnu.2011.07.007. Epub 2011 Aug 5. PMID 21820770
- [Derived] Klek S, Kulig J, Sierzega M, Szybinski P, Szczepanek K, Kubisz A, Kowalczyk T, Gach T, Pach R, Szczepanik AM. The impact of immunostimulating nutrition on infectious complications after upper gastrointestinal surgery: a prospective, randomized, clinical trial. Ann Surg. 2008 Aug;248(2):212-20. doi: 10.1097/SLA.0b013e318180a3c1. PMID 18650630